CLINICAL TRIAL: NCT01104311
Title: Multicenter Clinical Trial for Development of Guidelines of Adequate Blood Pressure Lowering in the Subacute Ischemic Stroke Patients Due to Intracranial Atherosclerosis
Brief Title: Strategy for Adequate Blood Pressure Lowering in the Patients With Intracranial Atherosclerosis
Acronym: STABLE-ICAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The enrollment was not done actively even though enrollment period was extended due to poor enrollment.
Sponsor: Asan Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Sun U. Kwon, department of neurology, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STABLE-ICAS
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Brain Ischemia
Keywords: Blood Pressure; Atherosclerosis; Brain Ischemia
MeSH Terms: conditions — Brain Ischemia; Atherosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aggressive BP lowering (Experimental): Lowering of systolic blood pressure between 110mmHg and 120mmHg during study period
  Interventions: Procedure: Aggressive BP lowering
- Modest BP lowering (Active Comparator): Lowering of systolic blood pressure between 130mmHg and 140mmHg
  Interventions: Procedure: modest blood pressure lowering

INTERVENTIONS:
Procedure: Aggressive BP lowering — adjust the amount and number of antihypertensive drugs to lowering of systolic blood pressure to target level
  Other Names: Aggressive BP control
  Arms: Aggressive BP lowering
Procedure: modest blood pressure lowering — adjust the amount and number of antihypertensive drugs
  Other Names: Modest BP control
  Arms: Modest BP lowering

SUMMARY:
To develop adequate blood pressure (BP) lowering strategy after subacute ischemic stroke patients with symptomatic severe intracranial atherosclerosis.

Primary hypothesis of this study is that aggressive BP control (lowering systolic BP between 110mmHg and 120mmHg) will not increase the ischemic lesion volumes in hemisphere compared to modest BP lowering (lowering systolic BP between 130mmHg and 140mmHg) in the patients with symptomatic severe intracranial atherosclerosis.

DETAILED DESCRIPTION:
The benefits of BP lowering in the prevention of primary and secondary prevention of stroke is established well, although absolute target BP level is uncertain. Current guidelines defined the normal BP as <120/80mmHg and recommend individualized target BP level.

Large well performed stroke prevention trials consistently showed that reduction of 10/5mmHg in patients with systolic BP below 140mmHg had clear benefits in the prevention of cardiovascular events. However, we have a dilemma about BP control in the patients with severe intracranial atherosclerosis.

Aggressive BP control will be more effective in the prevention of overall cardiovascular events than modest BP control, but aggressive BP control will reduce cerebral perfusion in the territory of severe intracranial disease and may increase the risk of ischemic damage.

The study will try to reveal aggressive BP control in the patients with symptomatic severe intracranial atherosclerosis is not increase ischemic lesion volume in hemisphere to compare modest BP control.

ELIGIBILITY:
Inclusion Criteria:

* acute symptomatic ischemic stroke having relevant lesion on DWI(Diffusion weighted image) MRI 7 days after and 42 days within onset.
* relevant stenosis(more than 50%) or occlusion from MCA(middle cerebral artery)(M1) to distal of ICA(internal carotid artery ) on MR(Magnetic resonance) angiogram or CT angiogram.
* mean systolic blood pressure>=140mmHg or taking antihypertensive drug on screening.

Exclusion Criteria:

* taking more than 3 antihypertensive drugs and mean systolic blood pressure>=150mmHg on screening.
* history of recent thrombolysis but stenosis or occlusion remained after thrombolysis.
* evidence of orthostatic hypotension
* suspicious embolic cerebrovascular stenosis
* planned state of cerebrovascular surgery or angioplasty or stent 7 months within screening.
* severe stroke-NIHSS>=16
* mean systolic blood pressure>=200mmHg which is not able to control on screening.
* abnormal blood test finding (abnormal LFT(liver function test), anemia, renal insufficiency)
* pregnant or breast-feeding
* severe stroke sequela or medical problem
* suspicious secondary hypertension
* disease causing edema or significant ankle edema on screening.
* severe heart failure which correspond to NYHA (New York Heart Association )heart failure classification class III or IV.
* inappropriate condition determined by investigator
* Patient who do not have FLAIR image on or two months prior to screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- South Korea (16):
  - Chungnam National University Hospital, Daejeon, Chungcheongnam-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Inje University Pusan Paik Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Eulji University Hospital, Daejeon
  - Kyungpook National University Hospital, Deagu
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Inchon
  - Dong-A University Hospital, Pusan
  - Kyung Hee University Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Eulji Hospital, Seoul
  - Boramae Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share data yet. It will be discussed with investigators who have been participating in this study.

REFERENCES:
- [Derived] Park JM, Kim BJ, Kwon SU, Hwang YH, Heo SH, Rha JH, Lee J, Park MS, Kim JT, Song HJ, Park JH, Yu S, Lee SJ, Park TH, Cha JK, Kwon HM, Kim EG, Lee SH, Lee JS, Lee J. Intensive blood pressure control may not be safe in subacute ischemic stroke by intracranial atherosclerosis: a result of randomized trial. J Hypertens. 2018 Sep;36(9):1936-1941. doi: 10.1097/HJH.0000000000001784. PMID 29847486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period of this study was from 07/Apr/2010 to 2/Apr/2014 and there had been recruited at medical clinic.
Pre-assignment Details: There were not any significant events and approaches for the overall study following participant enrollment.
Period: Overall Study
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Started | 66 | 66
Completed | 56 | 54
Not Completed | 10 | 12
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 2 | 2
Not completed — low compliance | 1 | 1
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participatns are analyzed by ITTpopulation ITT Population (Aggressive BP Lowring: 66, Modest BP Lowering: 63)
Groups:
- Aggressive BP Lowering: Lowering of systolic blood pressure between 110mmHg and 120mmHg during study period Aggressive BP lowering: adjust the amount and number of antihypertensive drugs to lowering of systolic blood pressure to target level
- Modest BP Lowering: Lowering of systolic blood pressure between 130mmHg and 140mmHg modest blood pressure lowering: adjust the amount and number of antihypertensive drugs
- Total: Total of all reporting groups
Arm/Group | Aggressive BP Lowering | Modest BP Lowering | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Customized [Mean (Standard Deviation); unit: years] | 64.8 (8.5) | 63.5 (11.2) | 64.2 (9.85)
Gender [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 41 | 36 | 77

OUTCOME MEASURES:

1. Primary Outcome: Ischemic Lesion Volume Change in the Whole Forebrain on Fluid Attenuation Inversion Recovery (FLAIR) Magnetic Resonance Imaging (MRI)
Description: The difference between final ischemic lesions volume and base ischemic lesions of both hemisphere on FLAIR MRI
Time Frame: Screening to 24 weeks
Population: The Number of Participants Analyzed by FAS(Full analysis)Population. FAS Population (Aggressive BP Lowering: 59, Modest BP Lowering: 52)
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Number analyzed (Participants) | 59 | 52
cc
  Screening | 11.2 (24.1) | 10.4 (19.4)
  Week 24 | 16.1 (39.3) | 12.6 (20.0)
  Change from Screening to Week 24 | 4.9 (18.3) | 2.2 (8.2)

2. Secondary Outcome: Change of the Ischemic Lesion Volume in Cerebral Hemisphere on FLAIR From Screening to Week 24 in FAS Population
Description: the difference between final ischemic lesions volume and base ischemic lesions in the territory of symptomatic intracranial disease on FLAIR MRI
Time Frame: 24 weeks
Population: The number of participants are analyzed by FAS population.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Number analyzed (Participants) | 59 | 52
cc
  Screening | 10.2 (22.6) | 9.9 (19.4)
  Week 24 | 15.0 (38.6) | 12.0 (20.0)
  Change from Screening to Week 24 | 4.9 (18.3) | 2.1 (8.2)

3. Secondary Outcome: The Number of Patients With New Ischemic Lesion in the Whole Forebrain on FLAIR MRI
Time Frame: 24 weeks
Population: The Number of Participants are analyzed by ITT (Intent to treat) Population. ITT Population (Aggressive BP Lowering: 66, Modest BP Lowering: 63)
Measure: Number; unit: participants
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Number analyzed (Participants) | 66 | 63
participants
  Yes | 10 | 5
  No | 49 | 47
  Missing data | 7 | 11

4. Secondary Outcome: Number of Participants With Cardiovascular Events From Screening to Week 24 in ITT Population.
Time Frame: 24 weeks
Population: The number of participants are analyzed by ITT Population.
Measure: Number; unit: participants
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Number analyzed (Participants) | 66 | 63
participants | 14 | 14

5. Secondary Outcome: Total Number of Cardiovascular Events Form Screening to Week 24 in ITT Population.
Time Frame: 24 Week
Population: The number of participants are analyzed by ITT population.
Measure: Number; unit: events
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Number analyzed (Participants) | 66 | 63
events | 17 | 15

6. Secondary Outcome: Number of Participants With Vascular Death From Screening to Week 24 in ITT Population.
Time Frame: 24 Weeks
Population: The number of participants are analyzed by ITT population.
Measure: Number; unit: participants
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Number analyzed (Participants) | 66 | 63
participants | 0 | 0

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: 24 Weeks
Population: The number of participants are analyzed by Safety population.
Measure: Number; unit: participants
Groups:
- Aggressive BP Lowering: Lowering of systolic blood pressure between 110mmHg and 120mmHg during study period
  Aggressive BP lowering: adjust the amount and number of antihypertensive drugs to lowering of systolic blood pressure to target level (Safety population: 65)
- Modest BP Lowering: Lowering of systolic blood pressure between 130mmHg and 140mmHg
  modest blood pressure lowering: adjust the amount and number of antihypertensive drugs (Safety population: 65)
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Number analyzed (Participants) | 65 | 65
participants
  With at least on AE | 51 | 47
  With at leat one SAE | 10 | 8
  Withdrawn due to AE | 1 | 4
  With AE due to the treatment | 5 | 3
  Who died | 0 | 0

ADVERSE EVENTS:
Arm/Group | Aggressive BP Lowering | Modest BP Lowering
Serious Adverse Events (participants affected / at risk) | 10/65 | 8/65
Other Adverse Events (participants affected / at risk) | 51/65 | 47/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive BP Lowering (N=65) | Modest BP Lowering (N=65)
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INFECTION BACTERIAL (Immune system disorders) | 1 (1) | 0 (0)
OVARIAN CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GENITAL NEOPLASM MALIGNANT MALE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PYELONEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
GASTRIC ULCER HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 1
STUPOR (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Vascular disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive BP Lowering (N=65) | Modest BP Lowering (N=65)
HEPATIC ENZYMES INCREASED (Hepatobiliary disorders) | 2 (2) | 2 (2)
GALLBLADDER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
BILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
SKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ROTARY CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERLIPAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
ABSCESS (Immune system disorders) | 0 (0) | 1 (1)
HERPES ZOSTER (Immune system disorders) | 1 (1) | 0 (0)
INFECTION BACTERIAL (Immune system disorders) | 1 (1) | 0 (0)
LEUCOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BLEPHARITIS (Eye disorders) | 1 (1) | 0 (0)
OVARIAN CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GENITAL NEOPLASM MALIGNANT MALE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSION AGGRAVATED (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION POSTURAL (Vascular disorders) | 1 (1) | 0 (0)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER CALCULUS (Renal and urinary disorders) | 1 (1) | 0 (0)
MICTURITION DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0)
MICTURITION FREQUENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
PYELONEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
FACE OEDEMA (Renal and urinary disorders) | 1 (1) | 1 (1)
AZOTAEMIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (3) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 2 (3)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (3)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
PERIODONTAL DISORDERS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PERIODONTAL DESTRUCTION (Gastrointestinal disorders) | 2 (2) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 1 (1)
C-REACTIVE PROTEIN INCREASED (General disorders) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 3 (3) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 4 (4)
ASTHENIA (General disorders) | 1 (1) | 2 (2)
ABDOMEN ENLARGED (General disorders) | 1 (1) | 0 (0)
SYNCOPE (General disorders) | 0 (0) | 1 (1)
ALLERGIC REACTION (General disorders) | 1 (1) | 0 (0)
FEVER (General disorders) | 2 (2) | 1 (1)
OEDEMA GENERALISED (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1)
AMNESIA (General disorders) | 0 (0) | 1 (1)
INSOMNIA (General disorders) | 2 (2) | 3 (3)
ANXIETY (General disorders) | 1 (1) | 1 (1)
DELIRIUM (General disorders) | 2 (2) | 0 (0)
ANOREXIA (General disorders) | 2 (2) | 1 (1)
DEPRESSION (General disorders) | 4 (4) | 5 (5)
PARAESTHESIA (Nervous system disorders) | 3 (3) | 2 (2)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 8 (10) | 12 (13)
PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (1)
DYSPHONIA (Nervous system disorders) | 0 (0) | 1 (1)
GAIT ABNORMAL (Nervous system disorders) | 1 (1) | 0 (0)
VISUAL FIELD DEFECT (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0)
PTOSIS (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 9 (9) | 11 (11)
SPEECH DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDERS (Nervous system disorders) | 1 (1) | 1 (1)
DEMENTIA (Nervous system disorders) | 0 (0) | 3 (3)
APRAXIA (Nervous system disorders) | 1 (1) | 0 (0)
STUPOR (Nervous system disorders) | 1 (1) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTITIS EXTERNA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS FUNGAL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Vascular disorders) | 1 (1) | 1 (1)
RENAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Vascular disorders) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PURPURA (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
COUGHING (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTIO (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No